CLINICAL TRIAL: NCT01639820
Title: Comparison of Pelvic Lymphadenectomy Versus Isolated Sentinel Lymph Node Biopsy Procedure for Early Stages of Cervical Cancers : a Randomized Multicenter Study With Evaluation of Medico-economic Impacts
Brief Title: Comparison of Pelvic Lymphadenectomy Versus Isolated Sentinel Lymph Node Biopsy Procedure for Early Stages of Cervical Cancers : a Multicenter Study With Evaluation of Medico-economic Impacts
Acronym: SENTICOL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008.515
Record Dates: First submitted 2010-09-07; First posted 2012-07-13 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Uterine Cervical Dysplasia
Keywords: Cervical cancer; early stage carcinoma; FIGO IA1 IA2 IB1 IIA; sentinel lymph node biopsy; pelvic lymphadenectomy; Surgery of uterine cervical carcinoma; medico economic impact; quality of life
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strategy A (Experimental): Only identification of sentinel nodes (without pelvic lymph-node dissection)
  Interventions: Procedure: only identification of sentinel nodes (without pelvic lymph-node dissection)
- Strategy B (Other): Identification of sentinel nodes + full pelvic lymph-node dissection
  Interventions: Procedure: identification of sentinel nodes + full pelvic lymph-node dissection

INTERVENTIONS:
Procedure: identification of sentinel nodes + full pelvic lymph-node dissection — identification of sentinel nodes + full pelvic lymph-node dissection
  Arms: Strategy B
Procedure: only identification of sentinel nodes (without pelvic lymph-node dissection) — only identification of sentinel nodes (without pelvic lymph-node dissection)
  Arms: Strategy A

SUMMARY:
Patients with early cervical cancer are usually treated with radical hysterectomy + pelvic lymph-node dissection. The study randomizes patients in 2 arms. The control arm is the classical surgical treatment including identification of the sentinel nodes, full pelvic lymph-node dissection and radical hysterectomy.

The experimental arm is only sentinel node identification + radical hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older,
* Absence of contraindication to laparoscopy,
* Uterine cervical carcinoma (every histological type except neuroendocrine),
* Stage IA1 with lymphatic tumor space involvement (LVSI) or IA2 diagnosed on cervical conization; or stage IA2, IB1 or IIA detected by clinical examination, confirmed by biopsy and measured by the MRI, the highest diameter being lower to 4 cm (a preoperative brachytherapy is allowed for tumors 2 to 4 cm in diameter),
* Negative pregnancy test for women able to procreate,
* Having the French National Social Security
* Signed informed consent

Exclusion Criteria:

* Neuroendocrine carcinoma,
* In situ carcinoma or stage IA1 without LVSI,
* Maximal tumoral diameter measured by MRI more than 4 cm,
* Stage IB1 by "down-staging",
* Stage IB2, IIB to IVB, including those who had a response to neoadjuvant treatment (chemotherapy or RT + chemotherapy) ,
* Presence of distant metastases,
* Progression of the cervical cancer or recurrence,
* History of pelvic lymphadenectomy,
* Other cancer diagnosed during the course of treatment,
* Contraindication to the injected products : allergy known to Patent Blue or rhenium sulfide,
* History of severe allergy (history of Quincke's edema, anaphylactic shock),
* Patient who does not understand, speak or write the French language,
* Pregnant woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with complications observed in the 2 arms during the per and post-operative period up to 6 months | 6 months after surgery

SECONDARY OUTCOMES:
Score of the questionnaire of quality of life at 30 days, 3 months and 6 months after surgery | 30 days, 3 months and 6 months after surgery
the costs of both studied strategies | At the surgery until 6 months
the detection rate of the sentinel node technique in the 2 arms | Day 1
the false negative rate in the control arm | Day 1
the sites of recurrence for each strategy | Day 1
Number of patients without 3 years-recurrence for each strategy | 3 years after surgery
Number of patient treated by radio chemotherapy because of the presence of micrometastases in the sentinel node | 30 days, 3 months and 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie, Hôpital Femme Mère Enfant, Bron, France

REFERENCES:
- [Result] Bats AS, Frati A, Mathevet P, Orliaguet I, Querleu D, Zerdoud S, Leblanc E, Gauthier H, Uzan C, Deandreis D, Darai E, Kerrou K, Marret H, Lenain E, Froissart M, Lecuru F. Contribution of lymphoscintigraphy to intraoperative sentinel lymph node detection in early cervical cancer: Analysis of the prospective multicenter SENTICOL cohort. Gynecol Oncol. 2015 May;137(2):264-9. doi: 10.1016/j.ygyno.2015.02.018. Epub 2015 Feb 26. PMID 25727652
- [Result] Mathevet P, Lecuru F, Uzan C, Boutitie F, Magaud L, Guyon F, Querleu D, Fourchotte V, Baron M, Bats AS; Senticol 2 group. Sentinel lymph node biopsy and morbidity outcomes in early cervical cancer: Results of a multicentre randomised trial (SENTICOL-2). Eur J Cancer. 2021 May;148:307-315. doi: 10.1016/j.ejca.2021.02.009. Epub 2021 Mar 24. PMID 33773275